CLINICAL TRIAL: NCT03957798
Title: Evaluation of a Motion-Activated Refusal-Skills Training Video Game for Prevention of Substance Use Disorder Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Maryland Treatment Centers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MREZ-001
Record Dates: First submitted 2019-04-16; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Relapse; Opioid Use; Marijuana Usage
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Treatment as Usual) (No Intervention): TAU consists of inpatient substance abuse treatment, followed by referral to outpatient treatment. For those who live within the outpatient geographic catchment area of the treatment center, patients are subsequently admitted to outpatient levels of care at treatment center. For the non-opioid population (primarily marijuana), this consists of the intensive outpatient program counseling sessions starting at a frequency of 3x/wk, tapering to 1x/wk with clinical progress with 12 wks target length of service. For the opioid population, this consists of a specialty youth opioid program with group and individual counseling, relapse prevention medications treatment, psychiatric assessment and treatment, also starting at a frequency of 3x/wk, tapering to 1x/wk with clinical progress, with indefinite target length of service. For those not within the outpatient geographic catchment area, patients are referred to local continuing care and outpatient levels of care convenient to their homes.
- Intervention (Treatment as usual + game) (Experimental)
  Interventions: Behavioral: RecoveryWarrior 2.0

INTERVENTIONS:
Behavioral: RecoveryWarrior 2.0 — RecoveryWarrior 2.0 was developed for use with Microsoft Kinect running on a Windows personal computer. All games made use of whole-body motion detection and the same voice-recognition feature. Body motions included a variety of arm, leg, and whole-body movements to physically enact the motions of destroying or evading images of drugs and drug paraphernalia. Voice features consisted of recognition of the refusal phrase "I'm Clean" Players could say or shout "I'm Clean" in order to gain additional strength for their game play avatar. All game art was created in a hyperrealistic, idealized, heroic style.
  Arms: Intervention (Treatment as usual + game)

SUMMARY:
The project proposes to continue the development of an intervention for relapse prevention in the form of a professional quality video game which rewards drug-rejecting physical motions and spoken refusal phrases. Phase I research findings showed that youth in recovery experienced increased low craving levels, strong levels of satisfaction, and interest in attending treatment sessions where the intervention is available - an important outcome since failure to attend treatment is highly correlated with relapse. In Phase II, the investigators propose to modify and expand the prototype based on customer feedback from treatment centers, counselors and patients. The investigators will test the effectiveness of the motion and voice-controlled game in a randomized controlled trial of youths in treatment for opioid use disorder who have access to the game for a month. The investigators will measure the effect of gameplay on successful completion of detoxification/inpatient treatment and rates of linkage to next level of outpatient treatment. The investigators will also measure the effect of gameplay compared to treatment as usual (TAU) during a subsequent episode of outpatient treatment (following inpatient), on rates of treatment attendance, treatment retention, urine drug test results, substance use self-report, treatment alliance, drug craving, and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* attending the MMTC inpatient program for primarily opioid or marijuana use disorder treatment
* ability to speak English

Exclusion Criteria:

* presence of a comorbid psychiatric condition that would make participation unsafe (eg, acute suicidality or unstable psychosis)
* pregnancy (because of the physical exertion required to play the game)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change in craving | baseline, discharge (up to 2 weeks from baseline), 4 week, 8 week
  For cravings, the 5-item Penn Alcohol Craving Scale was included at baseline, discharge, and postdischarge follow-up surveys, but modified to apply to marijuana and opioid use. It assessed the intensity of a participant's cravings (0=none at all to 6=very strong; sum of a maximum total of 30 points).
Change in self-efficacy | baseline, discharge (up to 2 weeks from baseline), 4 week, 8 week
  Self-efficacy for refusal of drugs was measured using the Marijuana Resistance Self-Efficacy scale at baseline, discharge, and follow-up surveys. It used a 4-item, 4-point scale (1=very easy to 4=very hard) that asked participants how easy or hard it would be to refuse the drug if offered and explain why they did not want it, why they wanted to avoid the situation in the first place, and why they wanted to leave the situation. It was adapted so that there was a similar version for opioid use. Participants were only asked about the primary drug for which they enrolled in treatment (ie, marijuana or opioids).

SECONDARY OUTCOMES:
Refusal Skill | 4 week
  Refusal skills were measured by asking participants if they agreed that they would use the phrase "I'm Clean" to refuse drugs (1=not agree to 5=highly agree), if they had used the phrase "I'm Clean" since discharge to refuse drugs, and if the phrase "I'm Clean" still rings in their head (not at all, less than once per week, a few times a week, or more often).
Abstinence of drug use | Baseline, 4 week, 8 week
  Participants were asked about the primary drug that they were in treatment for. Opioid and marijuana use at follow-up was ascertained by self-report of any use in the past 7 and 30 days.

OTHER OUTCOMES:
Counselor Alliance | discharge (up to 2 weeks from baseline), 4 week, 8 week
  Treatment rating was measured in three ways. First, it was measured with the Counselor Alliance Scale, which was taken from the Working Alliance Inventory, and used to measure treatment progress with the counselor at discharge, 4 weeks, and 8 weeks. The Counselor Alliance Scale uses 7-items and 7-points to measure how well participants believe counselors are working with them to improve their situation (1=never to 7=always).
Treatment Rating | 4 week, 8 week
  The treatment rating was also measured by asking participants about their satisfaction with inpatient care at the time of discharge and satisfaction with outpatient care at the 4-week and 8-week follow-up surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Greenberg, BFA, Principal Investigator — Media Rez LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abroms LC, Fishman M, Vo H, Chiang SC, Somerville V, Rakhmanov L, Ruggiero M, Greenberg D. A Motion-Activated Video Game for Prevention of Substance Use Disorder Relapse in Youth: Pilot Randomized Controlled Trial. JMIR Serious Games. 2019 May 23;7(2):e11716. doi: 10.2196/11716. PMID 31124471

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03957798/Prot_SAP_000.pdf